CLINICAL TRIAL: NCT02367716
Title: Post-market Study of Multi-Vector Left Ventricular Lead Performance in Chinese Patients With Chronic Heart Failure
Acronym: MVLV
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: SJM- CIP-CRD 733
Record Dates: First submitted 2015-02-12; First posted 2015-02-20 (Estimated); Results first posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: CRT — The study will include the Quartet™ family of left heart leads or any newer St. Jude Medical quadripolar CRT systems, including CRT-P systems, that China Food and Drug Administration (CFDA) might approve in the future

SUMMARY:
The purpose of this clinical study is to observe the safety and efficacy of the multi-vector left ventricular (LV) lead in Chinese patients that are indicated for Cardiac Resynchronization Therapy (CRT).

DETAILED DESCRIPTION:
This is a multi-center, non-randomized observational study.

The total duration of the study is expected to be 2.5 years. The clinical study will be conducted in no more than 15 centers in China. Approximately 120 subjects will be enrolled in this study. Subjects will be followed up at 3, 6, 12 months and every 6 months afterwards. All subjects need to be followed for at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Meets the current European Society of Cardiology (ESC) or American College of Cardiology Foundation (ACCF)/American Heart Association (AHA)/Heart Rhythm Society (HRS) Class I or Class IIa indications for CRT implant (including upgrades from single or dual chamber Implantable Cardioverter-Defibrillators (ICDs))
* Are ≥ 18 years of age at the time of enrolment.
* Are able to provide written Informed Consent prior to any study related procedure.

Exclusion Criteria:

* Patient who is unable to comply with the follow-up schedule.
* Patient who has any medical conditions that in the opinion of the investigator will not be appropriate to participate in the study .
* Patient has a life expectancy of less than 1 year due to any condition.
* Patients, who has a CRT device implanted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A patient meets the current ESC or ACCF/AHA/HRS Class I or Class IIa indications for CRT implant
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clay Cohorn, Study Director — Abbott
Locations (14):
- China (14):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The second Affliated hospital Anhui Medical University, Hefei, Anhui
  - The second Affiliated hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - The second hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing First Hospital Affiliated to Nanjing Medical University, Nanjing, Jiangsu
  - Zhejiang Greentown cardiovascular hospital, Hangzhou, Zhejiang
  - The First Affiliated hospital of Medical College of Zhejiang University, Hangzhou, Zhejiang
  - The second Affiliated hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Runrun Shaw Hospital College of Medicine Zhejiang University, Hangzhou, Zhejiang
  - Fuwai Hospital CAMS&PUMC, Beijing
  - Rui Jin hospital Shanghai Jiao Tong University School of Medicine, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm- St. Jude Medical Quartet™ LV Lead Model 1458Q: This post-market study was conducted as required by China FDA to characterize the safety and efficacy of the commercial St. Jude Medical (SJM) Quartet™ Left Ventricular (LV) lead model 1458Q implanted with any commercial SJM Unify Quadra CRT-D device or newer SJM quadripolar system (CRT-D or CRT-P).
  This is a single arm study.
  The first subject was enrolled on December 25, 2014 and the last subject was enrolled on March 25, 2016.
Period: Overall Study
Arm/Group | Treatment Arm- St. Jude Medical Quartet™ LV Lead Model 1458Q
Started | 121
Completed | 120
Not Completed | 1
Not completed — Patient did not meet inclusion criteria | 1

BASELINE CHARACTERISTICS:
Population: A total of 121 patients were recruited at 13 sites. However, one subject who was retrospectively enrolled after an existing implant did not meet inclusion criteria and therefore was not included in analyses as the subject was withdrawn by the investigator.
Groups:
- Treatment Arm: This post-market study was conducted as required by China FDA to characterize the safety and efficacy of the commercial SJM Quartet™ LV lead model 1458Q implanted with any commercial SJM Unify Quadra CRT-D device or newer SJM quadripolar system (CRT-D or CRT-P).
  This is a single arm study.
  The first subject was enrolled on December 25, 2014 and the last subject was enrolled on March 25, 2016.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: A total of 121 subjects were enrolled at 13 sites. However, one subject who was retrospectively enrolled after an existing implant did not meet inclusion criteria and therefore was not included in analyses as the subject was withdrawn by the investigator.
  years | 59.9 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: A total of 121 subjects were enrolled at 13 sites. However, one subject who was retrospectively enrolled after an existing implant did not meet inclusion criteria and therefore was not included in analyses as the subject was withdrawn by the investigator.
  Participants
    Female | 39
    Male | 81
New York Heart Association (NYHA) Class, n (%) [Count of Participants; unit: Participants] — Population: NYHA classification is determined by a physician and measures the severity of a patient's heart failure by evaluating heart failure symptoms and limitations. Class I patients have mild heart failure symptoms, while patients with Class IV have severe symptoms.
  Participants
    Class I | 1
    Class II | 38
    Class III | 63
    Class IV | 15
    Not Done | 3
Intrinsic QRS Duration [Mean (Standard Deviation); unit: milliseconds (ms)] — Population: A total of 113 patients had intrinsic QRS duration measured at baseline and are included in the analysis population.
  milliseconds (ms)
    number analyzed (Participants) | 113
    (all) | 158 (27.6)
Primary Cause of Cardiac Disease, n (%) [Count of Participants; unit: Participants] — Population: A total of 121 subjects were enrolled at 13 sites. However, one subject who was retrospectively enrolled after an existing implant did not meet inclusion criteria and therefore was not included in analyses as the subject was withdrawn by the investigator
  Participants
    Ischemic | 12
    Non-Ischemic | 108
Prior Cardiac Interventions, n (%) [Number; unit: participants] — Due to characters limitation for Row "PTCA/Stents/Atherectomy", the acronym "PTCA" stands for percutaneous transluminal coronary angiography. Population: A total of 121 subjects were enrolled at 13 sites. However, one subject who was retrospectively enrolled after an existing implant did not meet inclusion criteria and therefore was not included in analyses as the subject was withdrawn by the investigator
  participants
    Coronary Artery Bypass Graft | 0
    PTCA/Stents/Atherectomy | 9
Cardiac Medications, n (%) [Number; unit: participants] — Population: A total of 121 subjects were enrolled at 13 sites. However, one subject who was retrospectively enrolled after an existing implant did not meet inclusion criteria and therefore was not included in analyses as the subject was withdrawn by the investigator
  participants
    ACE Inhibitors | 73
    Adrenergics | 1
    Aldosterone Antagonist | 29
    Angiotensin Receptor Blocker | 29
    Anti-Arrhythmics | 31
    Anticoagulants | 8
    Antiplatelets | 37
    Beta Blockers | 87
    Calcium Channel Blockers | 5
    Cardiac Glycosides | 52
    Diuretics | 100
    Nitrates | 20
    Statins | 22
    Other | 51
    None | 6

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With LV Lead-related Serious Adverse Device Effects (SADEs)
Description: The primary safety endpoint is the number of participants with LV lead-related SADEs compared to the total number of analyzed participants.
Time Frame: From implantation to 6 months after implant procedure.
Population: Only subjects with data available for all evaluation time points (implant, pre-discharge, 3 months and 6 months) were considered evaluable and included in analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Arm of SJM Quartet™ LV Lead Model 1458Q: Enrolled in the treatment arm were patients implanted with the commercial SJM Quartet™ LV lead model 1458Q and any commercial SJM Unify Quadra CRT-D device or newer SJM quadripolar system (CRT-D or CRT-P).
Arm/Group | Treatment Arm of SJM Quartet™ LV Lead Model 1458Q
Number analyzed (Participants) | 120
Participants | 2

2. Secondary Outcome: The Number of Participants With Effective LV Pacing
Description: The effectiveness endpoint is the number of participants with effective LV pacing compared to the total number of analyzed participants. The following must be met to be considered effective LV pacing:
  * Pacing threshold (immediately after implant): for pacing threshold at a pulse width of 0.5 ms, the voltage must be ≤3.5 Voltage (V) in any LV lead vector.
  * Pacing stability (pre-discharge, 3 months and 6 months after implant): for pacing threshold at a pulse width of 0.5 ms, the voltage must be ≤6.0V in any LV lead vector.
  * Pacing impedance (immediately after implant): Impedance value in any LV lead vector must be in the normal range of 200-2000 ohm (Ω).
  * Table 9: Impedance stability (pre-discharge, 3 months and 6 months after implant): Impedance value in any LV lead vector must be in the normal range of 200-2000Ω.
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Arm of SJM Quartet™ LV Lead Model 1458Q: Enrolled in the treatment arm were patients implanted with the commercial SJM Quartet™ LV lead model 1458Q implanted and any commercial SJM Unify Quadra CRT-D device or newer SJM quadripolar system (CRT-D or CRT-P).
Arm/Group | Treatment Arm of SJM Quartet™ LV Lead Model 1458Q
Number analyzed (Participants) | 64
Participants | 48

3. Secondary Outcome: The Number of Participants in Each NYHA Functional Class
Description: This secondary objective is to count the number of participants in each NYHA functional class at 6 months; NYHA classification is determined by a physician and measures the severity of a patient's heart failure by evaluating heart failure symptoms and limitations. Class I patients have mild heart failure symptoms, while patients with Class IV have severe symptoms.
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm of SJM Quartet™ LV Lead Model 1458Q
Number analyzed (Participants) | 105
Participants
  NYHA Class I | 12
  NYHA Class II | 61
  NYHA Class III | 26
  NYHA Class IV | 3
  NYHA Not Done | 3

4. Secondary Outcome: The Intrinsic QRS Duration of Participants
Description: This secondary objective is to measure the intrinsic QRS duration of participants at 6 months.
Time Frame: 6 months
Population: Only subjects with data available for all evaluation time points (implant, pre-discharge, 3 months and 6 months) were considered evaluable and included in the analysis.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Treatment Arm of SJM Quartet™ LV Lead Model 1458Q
Number analyzed (Participants) | 76
Milliseconds | 141.9 (27.8)
Statistical Analysis 1: Comparison: Treatment Arm of SJM Quartet™ LV Lead Model 1458Q; Test type: Other — The mean change in QRS duration between Baseline and 6 months; Mean Difference (Final Values) = -13.9, Standard Deviation 29.6

ADVERSE EVENTS:
Time Frame: Safety surveillance of subjects started at enrollment and continued for at least 6 months post-enrollment for all subjects, unless the subject was withdrawn from the study or died prior to the 6-month visit. If a subject was retrospectively enrolled, the investigator reported any adverse events which occurred between the implant and the date of enrollment according to the protocol. Sites continued to collect adverse event data in subjects following the 6-month visit until the study completed.
Description: Clinical sites were required to report the following events to the Sponsor:
  * All Adverse Device Effects (ADEs), including procedure-related events
  * All Serious Adverse Devise Effects (SADEs) including procedure-related events
  * All deaths
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 3/120
Serious Adverse Events (participants affected / at risk) | 11/120
Other Adverse Events (participants affected / at risk) | 2/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=120)
Lead Dislodgement (Product Issues) | 3 (3) — Two events were lead dislodgments and are adjudicated as related to the Quartet™ 1458Q LV lead, other event are adjudicated as related to Right Ventricular (RV) Lead
Hematoma/Seroma (Product Issues) | 1 (1) — subject was diagnosed with pocket hematoma/seroma. This was treated by draining approximately 20ml of clear fluid from the pocket and the administration of prophylactic antibiotics.This event was related to PG
Inappropriate Shocks (Product Issues) | 4 (5) — inappropriate shock is the most frequently reported SADE, occurring in 3.3% (4/120) of enrolled subjects and none were due to the Quartet™ 1458Q LV lead. 4 events were related to Pulse Generator (PG). 1event was related to RV lead.
Infection (Infections and infestations) | 3 (3) — three events were assessed as a pocket infection,2 events were related to PG ,1event was related to system
Pneumothorax/Hemothorax (Injury, poisoning and procedural complications) | 1 (1) — chest x-ray showed that a pneumothorax had developed on the left side. The subject was successfully treated with closed thoracic drainage then discharged. This event was related to procedure
Rise in Threshold and Exit Block (Product Issues) | 1 (1) — This event was related to RV Lead
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=120)
Infection (Infections and infestations) | 1 (1) — One subject developed a pocket infection three days post-implant and was successfully treated with antibiotics. This event was related to PG
Pneumothorax/Hemothorax (Injury, poisoning and procedural complications) | 1 (1) — subject complained of breathing-related chest pain in the post-operative setting. A chest x-ray revealed left-sided pleural effusion, which was successfully treated by non-invasive means. This event was related to procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No